CLINICAL TRIAL: NCT01146574
Title: A Phase 2a, Multi-center, Randomized, Single Dose, Double-blind, Placebo-controlled Followed by a Multiple-dose, Single-blind, Placebo-controlled, Dose Escalation Study to Evaluate the Pharmacokinetics, Safety, Efficacy, Tolerability, and Pharmacodynamics of Sotatercept (ACE-011) for the Correction of Anemia in Subjects With End-stage Renal Disease (ESRD) on Hemodialysis (HD).
Brief Title: A Phase 2a Study To Evaluate The Pharmacokinetics, Safety, Efficacy, Tolerability, And Pharmacodynamics of Sotatercept (ACE-011) for the Correction of Anemia in Subjects With End-stage Renal Disease on Hemodialysis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ACE-011-REN-001
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Anemia
Keywords: End-Stage Renal Disease; Anemia; Hemodialysis; Renal Anemia; ESRD
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0.1mg/kg Sotatercept (Experimental): Approximately 8 subjects will be randomized to receive either a single 0.1 mg/kg subcutaneous dose of sotatercept or matching placebo in a 3:1 ratio
  Interventions: Biological: Sotatercept
- 0.3mg/kg Sotatercept (Experimental): Dose Group 1: 0.3 mg/kg sotatercept subcutaneous every 28 days
  Interventions: Biological: Sotatercept
- 0.5mg/kg Sotatercept (Experimental): Dose Group 2: 0.5 mg/kg sotatercept subcutaneous every 28 days
  Interventions: Biological: Sotatercept
- 0.7mg/kg Sotatercept (Experimental): Dose Group 3: 0.7 mg/kg sotatercept subcutaneous every 28 days
  Interventions: Biological: Sotatercept
- Placebo (Placebo Comparator): The Placebo to Sotatercept ratio is 1:3 meaning for every 1 patient that receives Placebo, 3 patients will receive Sotatercept.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Sotatercept — Part 1: Sotatercept single dose 0.1mg/kg subcutaneous Part 2: Sotatercept starting dose groups of 0.3mg/kg, 0.5mg/kg or 0.7 mg/kg in a sequential design, dosed subcutaneously every 28 days for up to 8 doses
  Other Names: ACE-011
  Arms: 0.1mg/kg Sotatercept; 0.3mg/kg Sotatercept; 0.5mg/kg Sotatercept; 0.7mg/kg Sotatercept
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is the first study in hemodialysis subjects with anemia to evaluate the pharmacokinetics, safety, efficacy, tolerability, and pharmacodynamics of sotatercept (ACE-011)

DETAILED DESCRIPTION:
Part 1:

Approximately 8 subjects will be randomized to receive either a single 0.1 mg/kg subcutaneous dose of sotatercept or matching placebo in a 3:1 ratio

Part 2:

Approximately 8 subjects will be randomized to each of the 3 sequential dose groups (0.3mg/kg or 0.5mg/kg or 0.7 mg/kg) with a 3:1 ratio of sotatercept or placebo (6 subjects in the sotatercept arm and 2 in the placebo arm). A total of 24-36 subjects may be randomized in the 3 dose groups.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥18 years of age.
* Subjects on hemodialysis for at least 12 weeks before screening
* Subjects on a stable dose of Erythrocyte Stimulating Agents product to maintain Hemoglobin (Hb) for at least 6 weeks prior to screening.
* 3 consecutive pre-dialysis Hb concentrations with a mean ≥10 to ≤ 12 g/dL (≥100 to ≤120 g/L) at screening and one pre-dialysis Hb concentration ≥8 to < 10 g/dL (≥ 80 to < 100 g/L) before randomization.
* Adequate iron status defined as serum transferrin saturation ≥ 20% before randomization.

Exclusion Criteria:

* Non renal causes of anemia.
* Subjects on peritoneal dialysis.
* Systemic hematological disease
* High sensitivity C-reactive protein >50mg/L at screening.
* Alanine transaminase (ALT) or aspartate transaminase (AST) laboratory values > 2 times the upper limit of normal (ULN) at screening.
* Uncontrolled diabetes mellitus (HbA1c > 9) at screening.
* Uncontrolled hypertension.
* Red Blood Count (RBC) transfusions within 8 weeks prior to screening.
* Active serious infection or history of recurrent serious infection likely to recur during the study
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product or to the iron products needed to normalize iron levels for subjects.
* Subjects that received treatment with another investigational drug or device within 28 days prior to Day 1
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2016-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Smith, MD, Study Director — Celgene Corporation
Locations (24):
- United States (24):
  - North American Research Institute, Azusa, California
  - West Glendale Dialysis, Glendale, California
  - California Institute of Renal Research, La Mesa, California
  - Academic Medical Center, Los Angeles, California
  - Academic Medical Research Institute, Los Angeles, California
  - Nephrology Specialist Medical Group, Orange, California
  - Pines Clinical Research Inc., Pembroke Pines, Florida
  - University of Kentucky, Lexington, Kentucky
  - Fresenius Medical Care North America MI, Kalamazoo, Michigan
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Nephrology and Hypertension Associates, LTD, Tupelo, Mississippi
  - St. Louis University Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Kidney Specialists of Southen Nevada, Las Vegas, Nevada
  - Brookview Hill Research Associates, LLC, Winston-Salem, North Carolina
  - MetroHealth Medical Systems, Cleveland, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Nephrology Associates, PC, Nashville, Tennessee
  - Corva Kidney Center Webster, Houston, Texas
  - Beechnut Dialysis Center, Houston, Texas
  - Miracle Medical Clinic, Houston, Texas
  - Gessner Dialysis Center, Houston, Texas
  - Tyler Nephrology Associates, PC, Tyler, Texas
  - University of Virginia at University Ave., Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1-Placebo: Participants received a single subcutaneous dose of placebo prior to dialysis on Day 1 via an IVRS.
- Part 1-ACE-011 0.1 mg/kg: Participants received a single subcutaneous dose of sotatercept (0.1 mg/kg) prior to dialysis on Day 1 via an IVRS
- Part 2- Placebo: Participants received a single subcutaneous dose of placebo
- Part 2-0.3 mg/kg: Participants received a single subcutaneous dose of 0.3 mg/kg sotatercept every 28 days for up to 8 doses
- Part 2-0.5 mg/kg: Participants received a single subcutaneous dose of 0.5 mg/kg sotatercept every 28 days for up to 8 doses
- Part 2-0.7 mg/kg: Participants received a single subcutaneous dose of 0.7 mg/kg sotatercept every 28 days for up to 8 doses
- Part 2-0.7/0.4 mg/kg: Participants received a subcutaneous dose of 0.7 mg/kg sotatercept loading followed by a subcutaneous dose of 0.4 mg/kg sotatercept every 14 days for up to 15 doses
Period: Overall Study
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Started | 1 | 6 | 11 | 9 | 8 | 9 | 6
Completed | 1 | 5 | 5 | 7 | 6 | 8 | 5
Not Completed | 0 | 1 | 6 | 2 | 2 | 1 | 1
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Other reasons | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Kidney transplant | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrew consent | 0 | 0 | 1 | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg | Total
Number analyzed (Participants) | 1 | 6 | 11 | 9 | 8 | 9 | 6 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 9 | 7 | 6 | 5 | 4 | 37
  >=65 years | 0 | 1 | 2 | 2 | 2 | 4 | 2 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 6 | 1 | 7 | 1 | 21
  Male | 0 | 5 | 7 | 3 | 7 | 2 | 5 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2 | 4 | 2 | 1 | 11
  Not Hispanic or Latino | 1 | 5 | 10 | 7 | 4 | 7 | 5 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 3 | 6 | 6 | 4 | 1 | 4 | 24
  White | 1 | 3 | 3 | 3 | 4 | 7 | 1 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Observed Maximum Concentration (Cmax)
Description: Cmax is a pharmacokinetic parameter defined as the observed maximum concentration of the study drug in the serum and/or blood. Cmax will be estimated from the sotatercept concentration versus time data using noncompartmental method.
Time Frame: From first dose up to Day 28
Population: Participants with evaluable pharmacokinetic data. Pharmacokinetic data was not recorded for participants who received placebo because no study drug was administered.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 9 | 8 | 9 | 6
ug/mL |  | 1.022 (0.576) |  | 2.40 (0.96) | 3.66 (0.67) | 3.97 (1.64) | 7.71 (1.97)

2. Primary Outcome: Time to Maximum Concentration (Tmax)
Description: Time to observed maximum concentration (Tmax) is defined as the amount of time in days for a drug to reach the maximum concentration after administration.
Time Frame: From first dose up to Day 28
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 9 | 8 | 9 | 6
Days |  | 6 [3 to 14] |  | 7 [3 to 14] | 8 [4 to 12] | 7 [4 to 10] | 5 [3 to 13]

3. Primary Outcome: Area Under Curve (AUC)-28 Days
Description: AUC-28 days is defined as area under the concentration-time curve over the first 28-day dosing interval
Time Frame: From first dose up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug·day/mL
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 9 | 8 | 9 | 5
ug·day/mL |  | 20.6 (11.4) |  | 50.64 (17.67) | 78.03 (13.34) | 87.51 (36.68) | 126.96 (20.75)

4. Primary Outcome: AUCinf: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity
Description: Area under the concentration-time curve from time zero extrapolated to infinity. Only Part 1 pharmacokinetic evaluable participants were pre-specified to be evaluated in this endpoint.
Time Frame: From first dose up to Day 28
Population: Pre-specified in the protocol to be collected in Part 1 pharmacokinetic evaluable participants only. Pharmacokinetic data was not recorded for participants who received placebo because no study drug was administered.
Measure: Mean (Standard Deviation); unit: ug·day/mL
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0 | 0
ug·day/mL |  | 35.8 (17.4) |  |  |  |  |

5. Primary Outcome: Apparent Total Clearance (CL/F)
Description: Apparent Total Clearance (CL/F) is defined as the volume of plasma from which the study drug is completely removed per unit of time. It is equal to the drug dose divided by the area-under-the-curve.
Time Frame: From first dose up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/day
Groups:
- Part 2-Placebo: Participants received a single subcutaneous dose of placebo
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2-Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 9 | 8 | 9 | 6
L/day |  | 3.22 (1.20) |  | 0.255 (0.068) | 0.261 (0.075) | 0.532 (0.654) | 0.298 (0.112)

6. Primary Outcome: Apparent Volume of Distribution Based on Terminal Phase (Vz/F)
Description: Apparent volume of distribution based on terminal phase (Vz/F) is defined as the apparent volume in which the current amount of drug in the body must be dispersed in order to give the current plasma concentration. Apparent volume of distribution is important for determining the dose required to produce a desired plasma concentration of the drug.
Time Frame: From first dose up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 0 | 0 | 0 | 0
mL/kg |  | 98 (38) |  |  |  |  |

7. Primary Outcome: Terminal Half-Life (t1/2,z)
Description: Terminal plasma half-life (t1/2,z) is the time taken for concentration of the study drug to decrease from its maximum concentration (Cmax) to half of Cmax in the blood plasma.
Time Frame: Days 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 15, 22, 29, 43, 57, 85 and 113
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 0 | 6 | 0 | 8 | 8 | 9 | 6
Day |  | 21.1 (3.9) |  | 24.3 (3.28) | 32.1 (19.9) | 22.2 (7.00) | 19.6 (2.91)

8. Secondary Outcome: The Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose up to 115 days post last dose
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 1 | 6 | 11 | 9 | 8 | 9 | 6
Participants | 1 | 6 | 7 | 8 | 6 | 8 | 4

9. Secondary Outcome: Number of Participants With Hemoglobin > 12g/dL
Description: Number of participants with hemoglobin > 12g/dL including Hb values obtained after first study drug dose and before any rescue.
Time Frame: Pre-dose; Dose 1-Days 1, 8, 15, 22, 29; Doses 2, 3, 4, 5, 6, 7-Days 1, 15, 29; Follow-up Phase Days 225, 253, 281, and 309
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 1 | 6 | 11 | 9 | 8 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 0

10. Secondary Outcome: Proportion of Participants With Rise in Hemoglobin > 2 g/dL During 4 Week Period
Description: Proportion of participants with rise in hemoglobin (Hb) > 2 g/dL during a 4-week period including Hb values obtained after first study drug dose and before any rescue.
Time Frame: as for outcome 9
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 1 | 6 | 11 | 9 | 8 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0

11. Secondary Outcome: Blood Pressure Changes From Baseline
Description: Blood pressure was generally recorded on the day of dialysis and represent pre-dialysis values. Baseline is defined as blood pressure measurements recorded on Day 1 of the first dose administered.
Time Frame: From pre-dose up to the final visit 112 days after last dose (up to 225 days)
Population: Safety population- all randomized participant who received at least 1 dose of sotatercept and had evaluable safety data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 1 | 6 | 9 | 9 | 8 | 9 | 6
mmHg
  Systolic Blood Pressure Baseline Day 1 | 151.0 (NA) — Standard deviation not calculated due to insufficient number of participants. | 142.8 (13.11) | 129.4 (27.99) | 145.9 (9.75) | 141.4 (18.72) | 139.9 (29.25) | 135.0 (25.09)
  Systolic Blood Pressure Final Visit: number analyzed (Participants) | 1 | 5 | 3 | 5 | 5 | 8 | 5
  Systolic Blood Pressure Final Visit | 163.0 (NA) — Standard deviation not calculated due to insufficient number of participants. | 134.6 (6.95) | 145.0 (26.91) | 167.0 (12.81) | 154.0 (34.47) | 154.3 (22.93) | 131.8 (12.79)
  Diastolic Blood Pressure Baseline Day 1 | 75.0 (NA) — Standard deviation not calculated due to insufficient number of participants. | 81.5 (7.56) | 71.6 (13.42) | 78.2 (12.45) | 74.3 (8.41) | 64.6 (13.33) | 72.0 (16.10)
  Diastolic Blood Pressure Final Visit: number analyzed (Participants) | 1 | 5 | 3 | 5 | 5 | 8 | 5
  Diastolic Blood Pressure Final Visit | 83.0 (NA) — Standard deviation not calculated due to insufficient number of participants. | 86.2 (15.93) | 79.7 (15.53) | 85.2 (9.83) | 83.6 (18.98) | 75.3 (9.19) | 71.6 (10.01)

12. Secondary Outcome: Changes in Follicle Stimulating Hormone (FSH)
Description: The change in follicle stimulating measured at pre-specified timepoints throughout the treatment period.
Time Frame: Day 1 (baseline), Day 15, Day 29, and Day 113
Population: All randomized participants in Part 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Part 1-Placebo | Part 1-ACE-011 0.1 mg/kg
Number analyzed (Participants) | 1 | 6
IU/L
  Day 1 (baseline) | 23.5 (NA) — Standard deviation not calculated due to insufficient number of participants | 36.9 (67.65)
  Day 15 | 17.1 (NA) — Standard deviation not calculated due to insufficient number of participants | 51.8 (80.76)
  Day 29 | 17.5 (NA) — Standard deviation not calculated due to insufficient number of participants | 37.4 (67.69)
  Day 113: number analyzed (Participants) | 1 | 5
  Day 113 | 11.8 (NA) — Standard deviation not calculated due to insufficient number of participants | 48.2 (78.81)

13. Secondary Outcome: Number of Participants With Hemoglobin > 10g/dL
Description: Number of participants with hemoglobin > 10g/dL including Hb values obtained after first study drug dose and before any rescue. Baseline is defined as hemoglobin measurements recorded on Day 1 of the first dose administered.
Time Frame: as for outcome 9
Population: All randomized participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 6
Participants | 3 | 3 | 5 | 7 | 2

14. Secondary Outcome: Number of Participants With Change From Baseline Hemoglobin ≥ 1g/dL
Description: Number of participants with a change from in hemoglobin values ≥ 1g/dL including Hb values obtained after first study drug dose and before any rescue. Baseline is defined as hemoglobin measurements recorded on Day 1 of the first dose administered.
Time Frame: as for outcome 9
Population: All randomized participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 6
Participants | 2 | 3 | 4 | 7 | 2

15. Secondary Outcome: Number of Participants With Hemoglobin > 10g/dL and Change From Baseline Hemoglobin ≥ 1g/dL
Description: Number of participants with Hemoglobin > 10g/dL and a change from in hemoglobin values ≥ 1g/dL including Hb values obtained after first study drug dose and before any rescue. Baseline is defined as hemoglobin measurements recorded on Day 1 of the first dose administered.
Time Frame: as for outcome 9
Population: All randomized participants in Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 6
Participants | 2 | 2 | 4 | 6 | 2

16. Secondary Outcome: Length of Time to Rescue Therapy
Description: The length of time in days that participants who were rescued received treatment. When applicable, participants were rescued for anemia. During the rescue, participants discontinued sotatercept and were unblinded to the study treatment. Participants who were rescued continued in the treatment phase of 200 days and a follow-up phase of 112 days after the treatment phase. Rescue is defined as the need for a blood transfusion or Erythropoiesis-stimulating agent (ESA) therapy.
Time Frame: From first dose up to blood transfusion or ESA therapy, up to approximately 209 days
Population: Participants in Part 2 who received rescue therapy
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 10 | 8 | 5 | 5 | 6
Days | 44.8 (43.96) | 69.8 (59.12) | 47.4 (32.86) | 100.4 (55.73) | 117.5 (73.37)

17. Secondary Outcome: Change From Baseline in Hemoglobin Values
Description: Dose Cycle 1 is defined as the first 28 days of treatment for Dose Groups 0.3 mg/kg, 0.5 mg/kg, and 0.7 mg/kg and the first 14 days of treatment for Dose Group 0.7/0.4 mg/kg. End of the Treatment Period is defined as the day before the follow-up phase started. Baseline is defined as hemoglobin measurements recorded on Day 1 of the first dose administered.
Time Frame: From first dose up to Day 225
Population: All randomized participants in Part 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part 2- Placebo | Part 2-0.3 mg/kg | Part 2-0.5 mg/kg | Part 2-0.7 mg/kg | Part 2-0.7/0.4 mg/kg
Number analyzed (Participants) | 11 | 9 | 8 | 9 | 6
g/L
  End of Dose Cycle 1: number analyzed (Participants) | 8 | 7 | 8 | 9 | 5
  End of Dose Cycle 1 | -3.3 (7.57) | -6.9 (6.94) | -2.9 (8.18) | 0.8 (5.85) | 1.0 (2.45)
  Peak Value During Dose Cycle 1: number analyzed (Participants) | 10 | 9 | 8 | 9 | 5
  Peak Value During Dose Cycle 1 | -0.9 (7.08) | 5.2 (8.24) | 7.1 (3.98) | 8.4 (3.75) | 5.4 (4.10)
  End of Treatment Period | 12.5 (12.42) | 12.8 (13.75) | 15.3 (8.22) | 15.0 (12.11) | 2.8 (6.91)

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 66 months). SAEs and Other AEs were assessed from first dose up to 115 days post last dose (up to 340 days).
Groups:
- Part 1 - Placebo: Participants received a single subcutaneous dose of placebo prior to dialysis on Day 1 via an IVRS.
- Part 1 - ACE-011 0.1 mg/kg: Participants received a single subcutaneous dose of sotatercept (0.1 mg/kg) prior to dialysis on Day 1 via an IVRS
- Part 2 - Placebo: Participants received a single subcutaneous dose of placebo
- Part 2 - 0.3 mg/kg: Participants received a single subcutaneous dose of 0.3 mg/kg sotatercept every 28 days for up to 8 doses
- Part 2 - 0.5 mg/kg: Participants received a single subcutaneous dose of 0.5 mg/kg sotatercept every 28 days for up to 8 doses
- Part 2 - 0.7 mg/kg: Participants received a single subcutaneous dose of 0.7 mg/kg sotatercept every 28 days for up to 8 doses
- Part 2 - 0.7/0.4 mg/kg: Participants received a subcutaneous dose of 0.7 mg/kg sotatercept loading followed by a subcutaneous dose of 0.4 mg/kg sotatercept every 14 days for up to 15 doses
Arm/Group | Part 1 - Placebo | Part 1 - ACE-011 0.1 mg/kg | Part 2 - Placebo | Part 2 - 0.3 mg/kg | Part 2 - 0.5 mg/kg | Part 2 - 0.7 mg/kg | Part 2 - 0.7/0.4 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/6 | 2/11 | 0/9 | 0/8 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/6 | 3/11 | 4/9 | 0/8 | 5/9 | 1/6
Other Adverse Events (participants affected / at risk) | 1/1 | 6/6 | 6/11 | 8/9 | 6/8 | 8/9 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Placebo (N=1) | Part 1 - ACE-011 0.1 mg/kg (N=6) | Part 2 - Placebo (N=11) | Part 2 - 0.3 mg/kg (N=9) | Part 2 - 0.5 mg/kg (N=8) | Part 2 - 0.7 mg/kg (N=9) | Part 2 - 0.7/0.4 mg/kg (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEART RATE IRREGULAR (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
TUMOUR THROMBOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 - Placebo (N=1) | Part 1 - ACE-011 0.1 mg/kg (N=6) | Part 2 - Placebo (N=11) | Part 2 - 0.3 mg/kg (N=9) | Part 2 - 0.5 mg/kg (N=8) | Part 2 - 0.7 mg/kg (N=9) | Part 2 - 0.7/0.4 mg/kg (N=6)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
VITREOUS HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 4 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
ASTHENIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 2
MEDICAL DEVICE COMPLICATION (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OEDEMA (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
PAIN (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ARTERIOVENOUS FISTULA SITE INFECTION (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CORNEAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TRACHEOBRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 1 | 0 | 0
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ARTERIOVENOUS GRAFT SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
EYE PENETRATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SKELETAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD PHOSPHORUS INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
EOSINOPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HEART RATE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VITAMIN D DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
CHROMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 3 | 0 | 4 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
STEAL SYNDROME (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
ORBITAL OEDEMA (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
CHILLS (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
ARTERIOVENOUS FISTULA SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.